CLINICAL TRIAL: NCT00372632
Title: Intermittent Preventive Treatment of Malaria With Sulfadoxine-Pyrimethamine in Different Zones of Drug Resistance in Rwanda
Brief Title: IPT of Malaria With SP in Different Zones of Drug Resistance in Rwanda
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Programme Nationale Lutte integré contre le Paludism, Ministère de la Santé
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 05 34 5 520
Record Dates: First submitted 2006-09-05; First posted 2006-09-07 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Non HIV Infected Pregnant Women
Keywords: Pregnancy malaria prevention
MeSH Terms: interventions — fanasil, pyrimethamine drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Drug: placebo
- sulfadoxine-pyrimethamine (Experimental)
  Interventions: Drug: Sulfadoxine-Pyrimethamine

INTERVENTIONS:
Drug: Sulfadoxine-Pyrimethamine — The intervention group receives 1500mg of sulfadoxine and 75mg of pyrimethamine at enrollment and in the third trimester.
  Other Names: fansidar
  Arms: sulfadoxine-pyrimethamine
Drug: placebo — The control group receives placebo similar in taste and appearance to to the experimental arm
  Arms: placebo

SUMMARY:
The present study will address the question whether the use of IPT using SP in pregnancy is efficacious in Rwanda, where it is going to be used for the first time, in areas with high levels of SP resistance. While the implementation of the new policy will take place in areas at low SP resistance level, where we expect pregnant women and newborns to benefit from it, it is of paramount importance to clarify which is the real impact of IPT/SPin areas of high SP drug resistance and at what level of SP resistance this strategy is still efficacious. As bed nets are a part of the actual control strategy of malaria in pregnancy all women will receive a bed net at enrolment

DETAILED DESCRIPTION:
The present study will address the question whether the use of IPT using SP in pregnancy is efficacious in Rwanda, where it is going to be used for the first time, in areas with high levels of SP resistance. While the implementation of the new policy will take place in areas at low SP resistance level, where we expect pregnant women and newborns to benefit from it, it is of paramount importance to clarify which is the real impact of IPT/SPin areas of high SP drug resistance and at what level of SP resistance this strategy is still efficacious. As bed nets are a part of the actual control strategy of malaria in pregnancy all women will receive a bed net at enrolment.

This will be a randomized blinded placebo controlled trial: women in the 16-28th week of gestation will be offered enrolment into the study and randomized to receive IPT/SP regimen or placebo once during the second and once in the third trimesters.

The study will be conducted in Mashesha (estimated SP drug resistance 20%, 12% in 2000), Kicukiro (40% SP resistance) and Rukara (60% SP resistance). In each of these sites there are about 1000 deliveries per year. According to DHMT data, over 75% of pregnant women attend antenatal clinics, usually booking between 15 and 25 weeks of gestation. Based on this study we expect to find placental malaria prevalence over 50% in all sites.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women between 16-28 weeks of gestation;
2. Residence within the catchment's area of the health facility;
3. Willing to deliver at the health facility;
4. Willing to ; adhere to all requirements of the study;
5. Willing to provide written informed consent;
6. Aged 21 years and above

Exclusion Criteria:

1. Severe anemia (Hb < 6 g/dL)
2. History of allergic reactions to sulfa drugs;
3. Taking other sulfa drugs as CTX;
4. History of known pregnancy complications (e.g. breech presentation, severe pre-eclampsia, prior caesarian section);
5. History or presence of major illnesses likely to influence pregnancy outcome including diabetes mellitus, severe renal or heart disease, or active tuberculosis, prior to randomization;
6. Any significant illness that requires hospitalization;
7. Intent to move out of the study catchment's area before delivery or deliver at relative's home out of the catchment's area;
8. Prior enrollment in the study or concurrent enrollment in another study

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1717 (Actual)
Dates: Start 2005-12; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
malaria infection will be defined as the presence of asexual stage parasites on thick smears made with maternal side placental blood and Maternal peripheral blood | maternal placental blood at delivery; maternal peripheral blood at monthly visits between 16 weeks of gestation and delivery

SECONDARY OUTCOMES:
LBW = birth weight <2,500 grams | at delivery
Premature delivery = delivery prior to 37 weeks gestation | at delivery
Spontaneous miscarriage = any spontaneous abortion before the end of gestation | at delivery
Stillbirth | at delivery
Cord blood parasitaemia = presence of asexual stage parasites in thick smears | at delivery
Neonatal death = infant death within the first 28 days of life | 7days and 6 weeks after delivery
Maternal anemia = Hb <11.0 g/dL | at monthly visits between 16 weeks of gestation and delivery
Maternal severe anemia = Hb <6 g/dL | at monthly visits between 16 weeks of gestation and delivery
Symptomatic maternal malaria infection = axillary temperature 37.5°C and asexual parasitaemia | at monthly visits between 16 weeks of gestation and delivery
Severe maternal adverse reactions to SP = severe cutaneous reactions (e.g., erythema multiform, Stevens-Johnson syndrome, or toxic epidermal necrolysis) | at monthly visits between 16 weeks of gestation and delivery plus at day 7 and week 6 after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Umberto D'Alessandro, MD,MSc, PHD, Study Director — Institute of Tropical Medicine Antwerp
Locations (1):
- Programme Nationale de Controle de Paludisms, Kigali, Rwanda